CLINICAL TRIAL: NCT00775125
Title: A Phase I, Open-label, Randomized, 2-way Crossover Trial in 40 Healthy Subjects to Investigate the Potential Pharmacokinetic Interactions Between Telaprevir and Darunavir/Ritonavir and Between Telaprevir and Fosamprenavir/Ritonavir at Steady-state.
Brief Title: VX-950-TiDP24-C124: A Phase I Trial to Investigate the Potential Pharmacokinetic Interactions Between Telaprevir and Darunavir/Ritonavir and Between Telaprevir and Fosamprenavir/Ritonavir at Steady-state.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec BVBA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR015208
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2010-12

CONDITIONS: Hepatitis C; Telaprevir; HIV
Keywords: VX-950-TiDP24-C124; VX-950-C124; HCV; DDI; telaprevir; darunavir; ritonavir; fosamprenavir; interaction; pharmacokinetics; steady-state
MeSH Terms: conditions — Hepatitis C | interventions — telaprevir; Darunavir; Ritonavir; fosamprenavir

INTERVENTIONS:
Drug: Telaprevir; Darunavir; Ritonavir; Fosamprenavir

SUMMARY:
The primary objectives are to determine the effect of steady-state DRV/rtv 600/100 mg twice daily (b.i.d.) on the steady-state pharmacokinetics of telaprevir 750 mg every (q) 8h and 1125 mg q12h and vice versa;- to determine the effect at steady-state of fAPV/rtv 700/100 mg b.i.d. on the steady-state pharmacokinetics of telaprevir 750 mg q8h and 1125 mg q 12h and vice versa; to determine the steady-state pharmacokinetics of telaprevir 750 mg q8h versus telaprevir 1125 mg q12h, alone and during coadministration of either steady-state DRV/rtv 600/100 mg b.i.d or fAPV/rtv 700/100 mg b.i.d.

DETAILED DESCRIPTION:
This is a Phase I, open-label, randomized (patients are assigned different treatments based on chance), 2-way crossover trial in 2 panels of healthy subjects to investigate the effect of steady-state darunavir/ritonavir (DRV/rtv) 600/100 mg b.i.d. (twice a day) or fosamprenavir/ritonavir (fAPV/rtv) 700/100 mg b.i.d. on the steady state pharmacokinetics (study of the bodily absorption, distribution, metabolism, and excretion of drugs) of telaprevir 750 mg q 8h and 1125 mg q12h, and vice versa.Telaprevir is being investigated for the treatment of HCV infection.The trial will enroll 40 subjects, divided over 2 panels of 20 subjects each. Subjects in Panel 1 will receive Treatments A and B, and subjects in Panel 2 will receive Treatments C and D, in a randomized order. In both panels, treatments will be separated by a washout period of at least 13 days. In Panel 1, Treatment A, subjects will receive telaprevir 750 mg q8h on Days 1 to 10, and telaprevir 1125 mg q12h on Days 11 to 13 with a morning dose on Day 14. In Panel 1, Treatment B, subjects will receive DRV/rtv 600/100 mg b.i.d. on Days 1 to 23, with an additional morning dose on Day 24, with coadministration of telaprevir 750 mg q8h on Days 11 to 20, and 1125 mg q12h on Days 21 to 23 with a morning dose on Day 24. In Panel 2, Treatment C, subjects will receive telaprevir 750 mg q 8h on Days 1 to 10, and telaprevir 1125 mg q12h on Days 11 to 13 with a morning dose on Day 14. In Panel 2, Treatment D, subjects will receive fAPV/rtv 700/100 mg b.i.d. on Days 1 to 23, with an additional morning dose on Day 24, with coadministration of telaprevir 750 mg q8h on Days 11 to 20, and 1125 mg q12h on Days 21 to 23 with a morning dose on Day 24. All intakes of study medication will be under fed conditions. Pharmacokinetic profiles of telaprevir and VRT-127394 (Rdiastereomer of telaprevir) will be measured up to 8 hours after intake of the morning dose on Day 10 of Treatments A and C and on Day 20 of Treatments B and D, and up to 12 hours after intake of the morning dose of Day 14 of Treatments A and C and on Day 24 of Treatments B and D. During Treatment B, pharmacokinetic profiles of DRV and ritonavir will be measured up to 12 hours after intake of the morning dose on Day 10, Day 20 and Day 24. During Treatment D, pharmacokinetic profiles of amprenavir and ritonavir will be measured up to 12 hours after intake of the morning dose on Day 10, Day 20 and Day 24. Safety and tolerability evaluations will be recorded at regular intervals throughout the trial period. Group A/C: telaprevir 750 mg each 8 hrs on Days 1-10, and telaprevir 1125 mg each 12hrs on Days 11-13 with a morning dose on Day 14. Group B: DRV/rtv 600/100 mg 2/day on Days 1-23 + morning dose on Day 24 + telaprevir 750 mg each 8 hrs on Days 11-20, and 1125 mg each 12hrs on Days 21 to 23 + morning dose on Day 24. Group D: fAPV/rtv 700/100 mg 2/day on Days 1-23 + morning dose on Day 24, + telaprevir 750 mg each 8hrs Days 11-20, and 1125 mg each 12hrs on Days 21-23 + morning dose on Day 24.

ELIGIBILITY:
Inclusion Criteria:

* Females in menopause for at least 3 years or surgically sterilized
* Nonsmoking or smoking no more than 10 cigarettes, or 2 cigars, or 2 pipes per day for at least 3 months prior to screening
* Normal weight at screening as defined by a body mass index (BMI) of 18 to 30 kg/m2, extremes included
* Able to comply with protocol requirements
* Healthy on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality and includes a physical examination, medical history, ECG, vital signs, and the results of blood biochemistry, blood coagulation and hematology tests and a urinalysis carried out at screening.

Exclusion Criteria:

* Subjects must not have a history of any illness that, in the opinion of the investigator or the subject's general practitioner, might confound the results of the study or pose an additional risk in administering trial drug(s) to the subject
* Subjects should currently not use prescription medication. Subjects should stop any short-duration courses of prescription medication at least 14 days before the screening visit. Potential subjects should not stop any chronic, prescribed medication being taken at the direction of a physician, without obtaining agreement from that physician
* Subjects should not have regular treatment with over-the-counter medications. Subjects should stop over-the-counter medications on the date of the screening visit but no less than 7 days prior to the first administration of study medication (Day 1 of Session I). Potential subjects should not stop any chronic, over-the-counter medication being taken at the direction of a physician, without obtaining agreement from that physician
* Subjects should not consumeherbal medications or dietary supplements and grapefruit or grapefruit juice, apple juice, or orange juice within 14 days before the first administration of study medication (Day 1 of Session I)
* Subjects should not have a history of drug or alcohol abuse or addiction within 2 years prior to dosing, or who test positive for alcohol or drugs such as amphetamine, barbiturates, benzodiazepines, cocaine, cannabinoids, opioids, metamphetamine and methadone during the screening period
* Subject should not have participated in a clinical study involving administration of an investigational drug within 3 months or 5 half lives (whichever is longer) prior to the screening visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Effect of steady-state DRV/rtv 600/100 mg b.i.d. and steady-state of fAPV/rtv 700/100 mg on the steady-state PK of telaprevir 750 mg q8h and 1125 mg q12h and vice versa. Steady-state PK on telaprevir 750 mg q8h and 1125 mg q12h alone.

SECONDARY OUTCOMES:
The secondary objective is to determine the short-term safety and tolerability of coadministration of telaprevir and DRV/rtv, and telaprevir and fAPV/rtv.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec-Virco Virology BVBA Clinical Trial, Study Director — Tibotec BVBA